CLINICAL TRIAL: NCT06617728
Title: Beyond the Quake: Exploring the Persistence of Phantom Limb Pain in Amputees from the 2023 Türkiye Earthquake
Brief Title: Phantom Limb Pain in Amputees After the 2023 Türkiye Earthquake
Status: Completed | Type: Observational
Sponsor: Mesut Bakır (Other)
Responsible Party: Sponsor-Investigator, Mesut Bakır, Clinical Professor, Mersin University
Organization: Mersin University (Other)
Other Study IDs: TURK-PLP-2023
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Phantom Limb Pain; Amputation; Pain Management; Earthquake
Keywords: Phantom Limb Pain; Amputation; Earthquake Injuries; Türkiye Earthquake 2023
MeSH Terms: conditions — Phantom Limb; Agnosia | interventions — Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Regional Analgesia Cohort: Participants receiving regional analgesia for pain management.
  Interventions: Procedure: Intervention 1: Regional Analgesia
- Group 2: Intravenous (IV) Analgesia Cohort: Participants receiving IV analgesia for pain management.
  Interventions: Drug: Intervention 2: Intravenous (IV) Analgesia

INTERVENTIONS:
Procedure: Intervention 1: Regional Analgesia — Regional analgesia techniques like epidural or peripheral nerve blocks.
  Groups: Group 1: Regional Analgesia Cohort
Drug: Intervention 2: Intravenous (IV) Analgesia — IV medications used for pain control, including opioids and non-opioid analgesics.
  Groups: Group 2: Intravenous (IV) Analgesia Cohort

SUMMARY:
The goal of this observational study is to investigate the prevalence and persistence of phantom limb pain (PLP) among amputees who experienced limb loss due to injuries sustained during the 2023 Türkiye earthquake. The main questions it aims to answer are:

What is the prevalence of phantom limb pain among earthquake-related amputees at different follow-up intervals? How do different pain management strategies, such as regional analgesia versus intravenous analgesia, affect the severity and persistence of phantom limb pain? Researchers will compare participants receiving regional analgesia to those receiving intravenous analgesia to see if regional techniques are associated with lower rates of phantom limb pain and improved quality of life.

Participants will:

Complete pain assessments using standardized questionnaires at 1 week, 3 months, 6 months, and 12 months post-amputation.

Provide information on their pain management experiences and the impact on their daily activities.

DETAILED DESCRIPTION:
This observational study aims to assess the prevalence, characteristics, and management of phantom limb pain (PLP) among individuals who underwent amputations due to injuries sustained during the 2023 Türkiye earthquake. Conducted at the Mersin University Pain Clinic, the study involves 39 patients who were followed for 12 months post-amputation. The primary focus is to evaluate how different analgesic methods, such as regional versus intravenous analgesia, influence the development and persistence of PLP and associated phantom limb sensations (PLS).

Patients were recruited from those treated at Mersin University Hospital immediately following the earthquake. Inclusion criteria included individuals aged 5 years and older who experienced amputation due to earthquake-related trauma. Exclusion criteria included pre-existing psychiatric disorders, history of neuropathic pain in the amputated limb, or inability to communicate due to cognitive impairment.

The study's primary outcomes are the prevalence of PLP and PLS at 1 week, 3 months, 6 months, and 12 months post-amputation. Pain intensity is measured using the Visual Analog Scale (VAS), and the impact of different analgesic techniques on pain severity and quality of life is analyzed. Secondary outcomes include the incidence of residual limb pain and the effectiveness of various pain management strategies in reducing pain symptoms over time.

This study is expected to contribute valuable insights into the management of PLP in disaster-related amputees, providing evidence to guide clinical practice and improve patient outcomes in similar post-disaster settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 5 years and older.
* Patients who have undergone amputation due to injuries sustained during the 2023 Türkiye earthquake.
* Experiencing phantom limb pain (PLP) as confirmed by a structured questionnaire.
* Able to provide informed consent or have consent provided by a legal guardian if under the age of 18.

Exclusion Criteria:

* Pre-existing psychiatric disorders that could interfere with pain perception or reporting.
* History of neuropathic pain in the amputated limb prior to the earthquake.
* Underwent surgical interventions in other parts of the body that may affect pain assessment.
* Inability to communicate effectively due to cognitive impairment or other medical conditions.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals who underwent amputations due to injuries sustained during the 2023 Türkiye earthquake. These patients were treated at the Pain Clinic of Mersin University Hospital and include both males and females aged 5 years and older. The study focuses on patients experiencing phantom limb pain (PLP) following amputation and evaluates the impact of different pain management strategies on their pain outcomes and quality of life. Participants include a diverse group with varying levels of amputation and injury severity, providing a comprehensive understanding of PLP in a post-disaster context.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of phantom limb pain | 1 week, 3 months, 6 months, and 12 months
  The percentage of amputee patients reporting PLP at each follow-up interval. PLP will be categorized as mild, moderate, or severe based on VAS scores.
o Prevalence of phantom limb sensations | 1 week, 3 months, 6 months, and 12 months
  The frequency of non-painful PLS such as tingling, itching, or movement sensations reported by patients at each follow-up period

SECONDARY OUTCOMES:
Incidence of residual limb pain | 1 week, 3 months, 6 months, and 12 months
  The number of patients reporting RLP at each follow-up interval, categorized based on VAS scores.
o Impact of Analgesic Methods | 1 week, 3 months, 6 months, and 12 months
  The effect of different analgesic methods on the prevalence and severity of PLP and PLS. Outcomes will be analyzed to determine which analgesic method is associated with lower pain scores and fewer phantom sensations.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Bakır, Assoc. Prof, Study Chair — Mersin University Faculty of Medicine, Pain Clinic
Locations (1):
- Mersin University Faculty of Medicine, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared upon reasonable request. Data will include demographic information, clinical outcomes, and responses to pain assessments. Researchers can request access by contacting the Principal Investigator at [mesutbakir@gmail.com]. Data will be available starting six months after publication of the primary results and for a period of five years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available starting six months after publication of the primary results and for a period of five years.
Access Criteria: De-identified participant data will be shared upon reasonable request. Data will include demographic information, clinical outcomes, and responses to pain assessments. Researchers can request access by contacting the Principal Investigator at [mesutbakir@gmail.com].